CLINICAL TRIAL: NCT00361673
Title: Reducing CVD (Cardiovascular Disease) Risk and Health Disparities Through Active Living Communities
Brief Title: Evaluating the Effect of Neighborhood Environments on Cardiovascular Risk Factors
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-0264; R21HL083866 (NIH); R21HL083866-01 (NIH)
Record Dates: First submitted 2006-08-04; First posted 2006-08-08 (Estimated); Last update posted 2013-12-25 (Estimated); Status verified 2013-12

CONDITIONS: Cardiovascular Diseases
Keywords: Health Disparities; Built Environments
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Cardiovascular disease (CVD) is one of the main causes of death in the United States. Research has shown that individuals who maintain an active lifestyle are less likely to develop CVD. This study will examine how neighborhood environments influence CVD risk factors of residents in and around the Stapleton community of Denver, Colorado.

DETAILED DESCRIPTION:
CVD is a major health problem in the United States. Individuals who live in an environment in which it is difficult to maintain an active lifestyle may be more at risk for developing CVD. Because of an increased interest in healthy living, urban planners and architects are now developing neighborhoods that are designed to encourage physical activity. Parks, walking and bicycle trails, wider sidewalks, and community recreation facilities are examples of amenities that are being included in these neighborhoods. By incorporating these enhancements, the Stapleton community in Denver, Colorado has been redeveloped as a more active living environment. The purpose of this study is to determine the effect of the neighborhood environment on the cardiovascular health of residents in five racially, ethnically, and socioeconomically diverse neighborhoods in or near the Stapleton community.

In Years 1 and 2 of this study, 200 households from each of the five neighborhoods will be randomly chosen to complete a survey regarding their cardiovascular health, physical activity level, and use and perception of their neighborhood environment and facilities, for a total of 1,000 surveys. Interviews and focus groups with members of the community will also be used to gather information. Additionally, a neighborhood council composed of community members will be formed to study disparities among the five neighborhoods in their use of their neighborhood environments, their physical activity levels, and their cardiovascular risk factors. In Year 2, study researchers will analyze the collected data and distribute the findings within the communities. They will also begin testing culturally and community relevant programs aimed at reducing CVD risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Live in one of the following five neighborhoods in the Greater Stapleton Community: Northeast Park Hill, Greater Park Hill, East Montclair, Stapleton, or Original Aurora
* Speak either English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of one of the following five neighborhoods in the Greater Stapleton Community: Northeast Park Hill, Greater Park Hill, East Montclair, Stapleton, or Original Aurora
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Actual)
Dates: Start 2006-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Effect of the neighborhood environment on the cardiovascular health of residents | Measured during Years 1 and 2 of the study

CONTACTS AND LOCATIONS:
Overall Officials: Debbi S. Main, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Denver, Aurora, Colorado
  - University of Colorado Denver, Denver, Colorado